CLINICAL TRIAL: NCT02348814
Title: Development of a Novel Biomarker for Liver Fibrosis
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Simon Beaven, Assistant Professor, University of California, Los Angeles
Other Study IDs: UL1TR000124-2016; UL1TR000124 (NIH)
Record Dates: First submitted 2015-01-14; First posted 2015-01-28 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Liver Fibrosis
Keywords: NAFLD, NASH
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimens include inflammatory markers (cytokines) and markers of metabolic dysfunction (adipokines):
  leptin, adiponectin, TNF-alpha, PAI-1, IL-6, MCP-1, and retinoids
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- normal weight: BMI 20-25
- overweight: BMI 25-30
- obese: BMI 30-35
- morbidly obese: BMI > 35
- non-diabetic: HgbA1c (<5.7%) and blood glucose (65-99 mg/dL) within normal range as defined at UCLA Clinical Lab
- diabetic: HgbA1c (>6.5%) and blood glucose (>100 mg/dL) as defined at UCLA Clinical Lab
- non-cirrhotic: Normal liver function tests (AST/SGOT, ALT, SGPT, alkaline phosphatase, bilirubin) as defined at UCLA Clinical Lab
- dyslipidemic: Abnormal lipid profile (Total cholesterol >170 mg/dL, LDL >100 mg/dL, HDL >130 mg/dL, triglycerides >150 mg/dL) as defined at UCLA Clinical Lab

SUMMARY:
The overall aim of this study is to validate a quantitative digital tool for staging liver fibrosis in biopsies from chronic human liver diseases and then evaluate it prospectively in patients.

DETAILED DESCRIPTION:
Preliminary data suggest that cholesterol and retinoid metabolism are tightly linked in these cells, prompting us to examine this relationship in the setting of obesity and diabetes. Specific aims have been developed to test the following hypotheses: 1) Quantifying liver fibrosis as a continuous variable will predict clinically significant outcomes in fatty liver disease related to metabolic syndrome; and 2) In a prospective cohort of patients, quantified liver fibrosis will correlate more strongly with tissue and circulating retinoid metabolites than with other, commonly measured serum markers.

This study offers a major innovation by performing accurate fibrosis quantification without any human intervention or post-analysis correction. In addition, we can test whether subtle differences in quantified fibrosis impact outcome for a given clinical stage of disease severity, possible because we are measuring fibrosis as a continuous variable, not a categorical one. We are using a disease-independent approach to evaluate anti-fibrotic agents in clinical trials and for evaluating other diagnostic markers.

We are also testing whether a novel diagnostic marker, retinoid storage, correlates with liver disease progression in humans. We propose to extend the study to address fatty liver disease, NAFLD/NASH, in the context of adult patients with abnormal liver tests, fatty liver identified on imaging, physical obesity, and diabetes. Clinical variables and outcomes to be recorded and analyzed include: morphology (age, gender, ethnicity, height, weight/BMI, waist circumference and steatosis on imaging studies); biochemistry (glucose intolerance or diabetes, complete blood counts, metabolic panels, liver function tests, cholesterol panels, insulin, and vitamin D levels); clinical outcomes (date of liver disease diagnosis and estimated duration of disease, listing on liver transplant list, occurrence of liver transplant or re-transplant, presence of cancer, and death); medications (current or previous prescribed, herbals, supplements taken for diabetes, dyslipidemia, hypertension, cardiovascular disease, or stroke); and disease exacerbation/modifying factors (presence of other chronic liver diseases such as NASH + HIV, liver toxins such as alcohol consumption, weight gain, or worsening diabetes).

Data will be collected from subjects who complete eight visits over a 24-month period. Assessments will include morphometric measurements, blood collection for laboratory analysis and completion of dietary history report.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* At least one liver function test abnormality (AST/SGOT, ALT/SOT, alkaline phosphatase, or bilirubin) defined as a value outside of the normal range at UCLA clinical labs. This must be present on at least two occasions within a 24 month consecutive period
* Any body mass index > 20
* One of the following:
* Clinical indication, according to standard of care assessment, for undergoing image-guided percutaneous (or transjugular) liver biopsy
* Eligible for weight loss (bariatric) surgery with fatty liver disease
* NAFLD/NASH patient who meets the above criteria and has already undergone a liver biopsy for diagnosis and disease staging
* NAFLD/NASH patient who meets above criteria but chooses not to participate in the liver biopsy, extra blood draws or the dietary assessment for the study.

Exclusion Criteria:

* Age < 18 years
* Current pregnancy
* Significant clinical co-morbidities that would preclude getting either a percutaneous or transjugular liver biopsy (i.e. platelets < 50, 000 or International Normalized Ratio (INR) > 1.5 or Hemoglobin < 8)
* Unwilling or unable to participate or consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects 18 years and older with at least one liver function test abnormality and body mass index > 20.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2019-01-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Composite of Clinical Outcomes-change over time | Participants will be followed up to 24 months; measured outcomes at 8 timepoints
  Date of liver disease diagnosis and estimated duration of disease, listing on liver transplant list, occurrence of liver transplant or re-transplant, presence of cancer (liver-related or otherwise), and death

SECONDARY OUTCOMES:
Composite of Morphometric Outcomes-change over time | Participants will be followed up to 24 months; measured outcomes at 8 timepoints
  height, weight (BMI), waist circumference, and steatosis (fat) on imaging studies

OTHER OUTCOMES:
Composite of Biochemical Outcomes-change over time | Participants will be followed up to 24 months; measured outcomes at 8 timepoints
  presence of glucose intolerance or diabetes, complete blood counts with differential, complete metabolic panels with liver function tests, cholesterol panels, insulin, C-reactive protein, vitamin D levels, and hepatocellular carcinoma or other solid tumor cancer markers

CONTACTS AND LOCATIONS:
Overall Officials: Simon Beaven, MD/PhD, Principal Investigator — UCLA Dept of Medicine, Division of Digestive Diseases
Locations (1):
- UCLA Clinical and Translational Research Center (CTRC), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No